CLINICAL TRIAL: NCT00893087
Title: Comparison of Pressure-, Flow- and NAVA-triggering in Pediatric and Neonatal Ventilatory Care
Brief Title: Comparison of Pressure-, Flow- and Neurally Adjusted Ventilatory Assistance (NAVA)-Triggering in Pediatric and Neonatal Ventilatory Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Tampere University (Other)
Responsible Party: Tero Kontiokari, MD, PhD, Associate Professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETTMK:122/2008
Record Dates: First submitted 2009-05-03; First posted 2009-05-05 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Respiration
Keywords: Ventilatory care, children, intensive care, asynchrony, triggering; Children needing ventilatory care
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Flow triggering
  Interventions: Device: Triggering mode of the ventilator; Device: Triggering method of the ventilator
- 2 (Active Comparator): Pressure triggering
  Interventions: Device: Triggering mode of the ventilator; Device: Triggering method of the ventilator
- 3 (Active Comparator): NAVA triggering
  Interventions: Device: Triggering mode of the ventilator; Device: Triggering method of the ventilator

INTERVENTIONS:
Device: Triggering mode of the ventilator — 10 min of each triggering mode
Device: Triggering method of the ventilator — Flow triggering
  Arms: 1
Device: Triggering method of the ventilator — Pressure triggering
  Arms: 2
Device: Triggering method of the ventilator — NAVA triggering
  Arms: 3

SUMMARY:
The purpose of this study is to study whether neurally adjusted ventilatory assist (NAVA) provides advantages over current methods in detecting patients own breathing efforts in pediatric and neonatal ventilatory care.

Our study hypothesis is that NAVA-technology is more accurate than currently used methods in detecting and assisting spontaneous breathing in children, and thus the patient-ventilator synchrony will improve.

DETAILED DESCRIPTION:
Asynchrony means that the timing of support given by the ventilator is different from patients own breathing pattern. Asynchrony during ventilatory care may increase the risk for complications, make the weaning more difficult and may affect the survival rates.

In this study we will compare two currently used methods pressure- and flow-triggering with a neurally adjusted ventilatory assist in synchronization of the ventilator support with patients own efforts.

ELIGIBILITY:
Inclusion Criteria:

* All children born over 30 weeks of gestation needing ventilatory care

Exclusion Criteria:

* Craniofacial malformation which does not allow feeding tobe positioning. Critical ventilatory or perfusion problems.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The time in ventilator-patient synchrony in each of the assist modes. | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Oulu, Oulu, Finland